CLINICAL TRIAL: NCT02074800
Title: A Phase 1, Randomized Study to Assess the Safety and Pharmacokinetics of a Single Intravenous Administration of CNTO 328 Derived From 2 Different Cell Lines in Healthy Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of a Single Intravenous Administration of CNTO 328 Derived From 2 Different Cell Lines in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR015271; C0328T08 (Other: Centocor)
Record Dates: First submitted 2014-02-27; First posted 2014-02-28 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Healthy; CNTO 328; Sp2/0-derived CNTO 328; CHO-derived CNTO 328; Safety; Pharmacokinetics
MeSH Terms: interventions — siltuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Participants will receive either 1.4 or 2.8 mg/kg of either Sp2/0-derived CNTO 328 or CHO-derived CNTO 328 or placebo.
  Interventions: Drug: CNTO 328 (Sp2/0-derived); Drug: CNTO 328 (CHO-derived); Drug: Placebo
- Part 2 (Experimental): Participants will receive 1.4 mg/kg of either Sp2/0-derived or CHO-derived CNTO 328.
  Interventions: Drug: CNTO 328 (Sp2/0-derived); Drug: CNTO 328 (CHO-derived)

INTERVENTIONS:
Drug: CNTO 328 (Sp2/0-derived) — Participants will receive a single-dose of Sp2/0-derived CNTO 328 intravenously (into the vein) either 1.4 or 2.8 mg/kg in Part 1 and 1.4 mg/kg in Part 2.
  Other Names: SILTUXIMAB
Drug: CNTO 328 (CHO-derived) — Participants will receive a single-dose of CHO-derived CNTO 328 intravenously (into the vein) either 1.4 or 2.8 mg/kg in Part 1 and 1.4 mg/kg in Part 2.
  Other Names: SILTUXIMAB
Drug: Placebo — Participants will receive a single-dose of matching placebo intravenously in Part 1.
  Arms: Part 1

SUMMARY:
The purpose of Part 1 of this study is to assess the safety and tolerability of 2 dose levels (1.4 and 2.8 mg/kg) of CHO-derived CNTO 328 and Sp2/0-derived CNTO 328. The purpose of Part 2 of this study is to access the pharmacokinetics (what the body does to the study medication) comparability of the 1.4 mg/kg dose of CHO-derived CNTO 328 and Sp2/0-derived CNTO 328.

DETAILED DESCRIPTION:
This is a single-dose and randomized (study medication is assigned by chance) study. This study will be conducted in 2 parts (Part 1 and Part 2). Approximately 144 participants will be enrolled in this study (24 participants in Part 1 and 120 participants in Part 2). Part 1 is the double-blind (neither physician nor participants know the treatment that the participant receives) and staggered parallel (a clinical study comparing the response in two or more groups of participants receiving different treatments) part of the study. Participants in Part 1 will receive either 1.4 or 2.8 mg/kg of either Sp2/0-derived CNTO 328 or CHO-derived CNTO 328 or placebo. Part 2 is the open-label (all people know the identity of the intervention) part of the study. Participants in Part 2 will receive 1.4 mg/kg of either Sp2/0-derived or CHO-derived CNTO 328. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored throughout the study. The total duration of study participation for each participant will be approximately 199 days including a screening phase (within 30 days before the first study medication administration) and a treatment phase (inpatient [hospitalization period] 12 days and outpatient [follow-up] visits up to 169 days).

ELIGIBILITY:
Inclusion Criteria:

* No clinically relevant abnormalities as determined by medical history, physical examination, blood parameters and having Body Mass Index (BMI) between 18.5 to 27 kg/m2 (BMI is calculated as weight [kilogram] divided by square of height [meter])
* Have an absolute neutrophil count of 2000 or more per cube millimeter at screening and one day before the study medication administration
* Agree to use adequate birth control measures for at least 100 days after study medication administration
* Agree not to use prescription medications (with the exception of hormonal contraceptives) within 14 days prior to study medication administration and through Day 85 of the study, unless approved by medical monitor
* Agree to limit caffeine/xanthine (eg, coffee, tea, chocolate, or caffeine-containing soft drinks) intake to less than 300 mg/day through Day 85 of the study

Exclusion Criteria:

* Have a current or past history of disease or dysfunction of the pulmonary, cardiovascular, endocrine, hematologic, neurological, immune, gastrointestinal, genitourinary, or other body system, that is clinically significant in the opinion of the investigator
* Have a current or past history of thrombocytopenia (a low platelet count) or bleeding abnormality or elevations in triglycerides that require treatment
* Have evidence of any chronic medical condition requiring prescription medications (eg, hypertension, elevated cholesterol/triglycerides, asthma, or diabetes)
* Positive serology test for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at screening
* Positive urine toxicology screen and substances of abuse, including but not limited to alcohol, cocaine, cannabinoids, phencyclidine, amphetamines, benzodiazepines, barbiturates, opiates, propoxyphene, and methadone

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability in Part 1 | Up to Day 199
Maximum observed serum concentration (Cmax) of CNTO 328 in Part 2 | Day 1 (predose, end of infusion, and postdose at Hours 1, 2, 4, and 8), Days 2 to 6, and Days 8, 15, 22, 29, 36, 43, 50, 71, and 85
  This sample will be used for pharmacokinetics analysis. Cmax is defined as the maximum observed analyte concentration.
Area under the serum concentration-time curve from Day 0 to Day 84 (AUC 0-84D) of CNTO 328 in Part 2 | Day 1 (predose, end of infusion, and postdose at Hours 1, 2, 4, and 8), Days 2 to 6, and Days 8, 15, 22, 29, 36, 43, 50, 71, and 85
  This sample will be used for pharmacokinetics analysis. AUC 0-84D is a measure of the serum concentration of the study medication over time. It is used to characterize drug absorption.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability in Part 2 | Up to Day 199
Immune response of CNTO 328 in Part 1 and Part 2 | Day 1 (predose), Days 85, 113, and 169
  Immune response will be evaluated by analyzing serum samples for the determination of the presence of antibodies to CNTO 328.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Clinical Trial, Study Director — Centocor, Inc.
Locations (2):
- United States (2):
  - Lincoln, Nebraska
  - Neptune City, New Jersey